CLINICAL TRIAL: NCT05148481
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of BIIB104 in Healthy Japanese and Non-Japanese Participants
Brief Title: A Study to Evaluate Safety and Pharmacokinetics of BIIB104 in Healthy Japanese and Non-Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 263HV108
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BIIB104: Dose 1 (Experimental): Japanese and non-Japanese participants will receive BIIB104, Dose 1, oral capsule, BID, from Day 1 through Day 9 with an additional dose on Day 10.
  Interventions: Drug: BIIB104
- BIIB104: Dose 2 (Experimental): Japanese and non-Japanese participants will receive BIIB104, Dose 2, oral capsule, BID, from Day 1 through Day 9 with an additional dose on Day 10.
  Interventions: Drug: BIIB104
- Placebo (Placebo Comparator): Japanese and non-Japanese participants will receive BIIB104-matching placebo, oral capsule, BID, from Day 1 through Day 9 with an additional dose on Day 10.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB104 — Administered as specified in the treatment arm
  Arms: BIIB104: Dose 1; BIIB104: Dose 2
Drug: Placebo — Administered as specified in the treatment arm
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the pharmacokinetics (PK) of BIIB104 in healthy Japanese and non-Japanese participants. The secondary objective of the study is to evaluate the safety and tolerability of multiple, oral doses of BIIB104 administered twice daily (BID) for 9 days, with an additional dose occurring in the morning on Day 10 in healthy Japanese and non-Japanese participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a body mass index between 18 and 30 kilograms per meter square (kg/m^2), inclusive, and total body weight >50 kilograms (kg) [110 pounds (lb)].
* For Japanese participants, was born in Japan, and biological parents and grandparents were of Japanese origin.
* For Japanese participants, if living outside Japan for more than 5 years, must not have significantly modified diet since leaving Japan.
* Non-Japanese participants must have a screening weight within ±20% of the mean value for Japanese participants.

Key Exclusion Criteria:

* Participation in other studies involving treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to randomization and/or during study participation.
* History of severe allergic or anaphylactic reactions, systemic hypersensitivity reaction to BIIB104, or any allergic reactions that in the opinion of the investigator are likely to be exacerbated by any component of the study treatment.
* History of seizures or a condition with risk of seizures.
* History of, or positive test result at Screening for, human immunodeficiency virus (HIV).
* Chronic, recurrent, or serious infection, as determined by the investigator, within 6 months prior to screening or between screening and Day 1.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 31 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of BIIB104 | Up to Day 11
Time to Reach Maximum Observed Concentration (Tmax) of BIIB104 | Up to Day 11
Area Under the Concentration-Time Curve Within a Dosing Interval for Single Dose [AUC(tau,sd)] of BIIB104 | Up to Day 11
Maximum Observed Concentration at Steady State (Cmax,ss) of BIIB104 | Up to Day 11
Time to Reach Maximum Observed Concentration at Steady State (Tmax,ss) of BIIB104 | Up to Day 11
Area Under the Concentration-Time Curve Over a Uniform Dosing Interval Tau at Steady State [AUC(tau,ss)] of BIIB104 | Up to Day 11
Apparent Total Body Clearance (CL/F) of BIIB104 | Up to Day 11
Apparent Volume of Distribution (Vz/F) of BIIB104 | Up to Day 11
Elimination Half-Life (t½) of BIIB104 | Up to Day 11
Accumulation Ratio for Steady State of BIIB104 | Up to Day 11
  Accumulation ratio for steady state is defined as area under the concentration-time curve over a uniform dosing interval tau at steady state divided by area under the concentration-time curve within a dosing interval for single dose [AUC(tau,ss)/AUC(tau,sd)].
Trough Concentration (Ctrough) of BIIB104 | Up to Day 11

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Day 1 up to Day 25
  An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Number of Participants with Serious Adverse Events (SAEs) | From screening up to Day 25
  A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, in the view of the investigator, places the participant at immediate risk of death (a life-threatening event), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect or is a medically important event.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/